CLINICAL TRIAL: NCT01785472
Title: A Multi-center, Randomized, Double-blind, Active-controlled, 8-week Study to Evaluate the Efficacy and Safety of LCZ696 in Comparison to Olmesartan in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of LCZ696 in Comparison to Olmesartan in Asian Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696A2315; CLCZ696A2315 (Other: Novartis)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; LCZ696
MeSH Terms: conditions — Essential Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; olmesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LCZ696 200 mg (Experimental): Patients will be treated with one LCZ696 200 mg tablet and one placebo of LCZ696 once daily(qd) for eight weeks along with placebo of Olmesartan 20 mg capsule once daily.
  Interventions: Drug: LCZ696; Drug: Placebo of LCZ696; Drug: Placebo of Olmesartan
- LCZ696 400 mg (Experimental): Patients will start with one LCZ696 200 mg tablet and one placebo of LCZ696 once daily (qd) for one week, thereafter all patients in the treatment group will be up-titrated to two LCZ696 200 mg tablets (400 mg of LCZ696) qd for the remaining seven weeks. Placebo of Olmesartan 20 mg capsule once daily also will be taken.
  Interventions: Drug: LCZ696; Drug: Placebo of LCZ696; Drug: Placebo of Olmesartan
- Olmesartan 20 mg (Active Comparator): Patients will be treated with Olmesartan 20 mg for eight weeks once daily along with placebo of LCZ696 tablets once daily.
  Interventions: Drug: Olmesartan; Drug: Placebo of LCZ696

INTERVENTIONS:
Drug: LCZ696 — LCZ696 200 mg tablet
  Arms: LCZ696 200 mg; LCZ696 400 mg
Drug: Olmesartan — Olmesartan 20 mg capsule
  Arms: Olmesartan 20 mg
Drug: Placebo of LCZ696 — Placebo tablet of LCZ696 200 mg once daily
Drug: Placebo of Olmesartan — Placebo capsule of olmesartan 20 mg once daily
  Arms: LCZ696 200 mg; LCZ696 400 mg

SUMMARY:
This study will assess the efficacy and safety of multiple doses of LCZ696 compared to olmesartan in Asian patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild-to-moderate hypertension, untreated or currently taking antihypertensive therapy.
* Treated patients (using antihypertensive treatments within 4 weeks prior to Visit 1) must have an msSBP≥150 mmHg and <180 mmHg at the randomization visit (Visit 201) and msSBP≥140 mmHg <180 mmHg at the visit immediately preceding Visit 201 (Visit 102 or 103).
* Untreated patients (newly diagnosed with essential hypertension or having a history of hypertension but have not been taking any antihypertensive drugs for at least 4 weeks prior to Visit 1) must have an msSBP≥150 mmHg and <180 mmHg at both Visit 1 and Visit 201.
* Patients must have an absolute difference of ≤15 mmHg in msSBP between Visit 201 and the immediately preceding visit.

Exclusion Criteria:

* Patients with severe hypertension (msDBP ≥110 mmHg and or msSBP ≥180 mmHg).
* History of angioedema, drug-related or otherwise, as reported by the patient.
* History or evidence of a secondary form of hypertension, including but not limited to any of the following: renal parenchymal hypertension, renovascular hypertension (unilateral or bilateral renal artery stenosis), coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, pheochromocytoma, polycystic kidney disease, and drug-induced hypertension.
* Patients who previously entered a LCZ696 study and had been randomized or enrolled into the active drug treatment epoch.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1438 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (39):
- China (21):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Fuzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- Philippines (2):
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Quezon City
- Novartis Investigative Site, Singapore, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Koyang, Kyunggi
- Taiwan (8):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei County, Taiwan
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Douliu
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taipei
- Thailand (4):
  - Novartis Investigative Site, Rajathevee, Thailand
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Started | 479 | 473 | 486
Full Analysis Set (FAS) | 479 | 472 | 484
Safety Set (SAF) | 478 | 472 | 484
Completed | 455 | 454 | 464
Not Completed | 24 | 19 | 22
Not completed — Adverse Event | 5 | 4 | 6
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Protocol deviation | 0 | 2 | 2
Not completed — Subject/guardian decision | 15 | 10 | 11
Not completed — Technical problems | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All patients who were randomized. Patients were analyzed according to the treatment they were assigned to at the randomization. However, patients who were not qualified for randomization and were inadvertently randomized into the study were excluded from the FAS, provided these patients did not receive study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg | Total
Number analyzed (Participants) | 479 | 472 | 484 | 1435
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (10.17) | 58.1 (9.71) | 57.4 (10.14) | 57.7 (10.01)
Gender [Count of Participants; unit: Participants]
  Female | 227 | 229 | 223 | 679
  Male | 252 | 243 | 261 | 756

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) Between LCZ696 200 mg Versus Olmesartan 20 mg
Description: Sitting BP measurements will be performed at screening through end of study at every visit. Four separate sitting BP measurements will be obtained with a full two minute interval between measurements.
Time Frame: baseline, 8 weeks
Population: Only participants, who had both baseline and week 8 values, were included in the analysis. The FAS included all randomized participants who received study medication and had post baseline BP assessments
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 477 | 479
mmHg | -20.48 (0.61) | -18.15 (0.61)
Statistical Analysis 1: Comparison: LCZ696 200 mg vs Olmesartan 20 mg; Test type: Non-Inferiority or Equivalence — The statistical test was made at a one-sided significance level of 0.025; p < 0.001, ANCOVA; least Square Means net difference = -2.33, 95% CI [-4.00 to -0.66], Standard Error of Mean 0.85

2. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) Between LCZ696 400 mg Versus Olmesartan 20 mg
Description: as for outcome 1
Time Frame: baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 469 | 479
mmHg | -21.67 (0.62) | -18.15 (0.61)

3. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP) Between LCZ696 200, and LCZ696 400 mg Versus Olmesartan 20 mg
Description: Sitting BP measurements were performed at screening through the end of the study at every study visit. A negative change from baseline indicates improvement
Time Frame: baseline, 8 weeks
Population: Participants from the full analysis set (FAS), who had both baseline and week 8 values, were included in the analysis. The FAS included all participants who received study medication and had post baseline BP assessments
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 477 | 469 | 479
mmHg | -8.10 (0.37) | -8.80 (0.38) | -6.86 (0.37)

4. Secondary Outcome: Change From Baseline in Office Pulse Pressure (msPP)
Description: Four separate sitting BP measurements should be obtained with a full two minute interval between measurements.
Time Frame: baseline, 8 weeks
Population: Participants from the full analysis set (FAS), who had both baseline and endpoint were included in the analysis. The FAS included all participants who received study medication and had post baseline BP assessments
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 477 | 469 | 479
mmHg | -12.35 (0.42) | -12.93 (0.43) | -11.25 (0.42)

5. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Blood Pressure
Description: In this analysis, mean 24 hour ambulatory systolic blood pressure maSBP, mean 24 hour ambulatory diastolic blood pressure maDBP, daytime and nightime maSBP and maDBP will be reported. Ambulatory blood pressure monitoring over a 24 hour period will be conducted at two time points during the study.
Time Frame: baseline, 8 weeks
Population: A subset of participants, who participated in ambulatory blood pressure monitoring, was analyzed
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 184 | 182
mmHg
  maSBP | -12.07 (0.49) | -12.76 (0.49) | -10.26 (0.49)
  maDBP | -6.36 (0.31) | -6.82 (0.31) | -5.61 (0.31)

6. Secondary Outcome: Sub-group Analysis for Change From Baseline in Mean Ambulatory Systolic Blood Pressure in Dippers.
Description: Twenty four hour ABPM was performed twice duirng the study at baseline and week 8. The second ABPM assessment was performed only in participants who had successfully completed the ABPM assessment at baseline. Dippers were defined as participants who showed a decrease of at least 10% in maSBP during the night (10pm-6am) compared with the daytime level. A negative change from baseline indicates improvement
Time Frame: baseline, 8 weeks
Population: A subset of participants, who participated in ambulatory blood pressure monitoring, was analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 55 | 79 | 74
mmHg
  Hour 1 | -13.22 (16.506) | -15.02 (14.578) | -9.07 (17.597)
  Hour 2 | -17.24 (20.423) | -18.11 (15.343) | -13.95 (19.247)
  Hour 3 | -14.99 (19.378) | -16.83 (16.312) | -14.51 (18.436)
  Hour 4 | -13.09 (19.460) | -16.37 (18.710) | -14.63 (18.824)
  Hour 5 | -11.19 (19.376) | -18.88 (16.636) | -14.64 (21.177)
  Hour 6 | -13.66 (16.785) | -19.19 (17.771) | -11.54 (21.885)
  Hour 7 | -11.74 (21.552) | -18.07 (19.748) | -11.74 (24.674)
  Hour 8 | -13.84 (17.365) | -16.12 (16.696) | -12.99 (20.555)
  Hour 9 | -16.33 (16.437) | -15.64 (18.915) | -13.33 (18.360)
  Hour 10 | -13.81 (17.670) | 15.13 (18.014) | -10.89 (19.814)
  Hour 11 | -12.98 (16.856) | -15.93 (19.022) | -7.66 (18.816)
  Hour 12 | -8.99 (17.913) | -15.54 (20.397) | -10.51 (19.516)
  Hour 13 | -12.46 (18.694) | -13.28 (17.014) | -11.49 (18.587)
  Hour 14 | -9.64 (17.001) | -12.33 (16.449) | -6.66 (17.906)
  Hour 15 | -7.73 (17.362) | -10.12 (14.433) | -7.81 (15.383)
  Hour 16 | -4.92 (14.788) | -12.82 (13.386) | -4.40 (15.974)
  Hour 17 | -10.20 (15.780) | -12.43 (14.397) | -7.19 (14.937)
  Hour 18 | -9.84 (15.789) | -11.70 (13.799) | -8.90 (14.907)
  Hour 19 | -8.94 (12.283) | -12.20 (15.012) | -5.76 (16.029)
  Hour 20 | -8.03 (19.411) | -15.04 (14.647) | -4.83 (15.953)
  Hour 21 | -9.47 (16.984) | -14.33 (13.585) | -9.97 (16.552)
  Hour 22 | -12.62 (17.527) | -17.20 (14.304) | -9.95 (18.490)
  Hour 23 | -9.23 (20.068) | -16.63 (15.752) | -14.09 (25.454)
  Hour 24 | -8.43 (15.330) | -15.76 (17.392) | -12.71 (15.199)

7. Secondary Outcome: Sub-group Analysis for Change From Baseline in Mean Ambulatory Diastolic Blood Pressure in Dippers.
Description: as for outcome 6
Time Frame: baseline, 8 weeks
Population: A subset of participants, who participated in ambulatory blood pressure monitoring, was analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 55 | 79 | 74
mmHg
  Hour 1 | -7.93 (10.377) | -7.38 (8.786) | -5.99 (11.811)
  Hour 2 | -8.47 (12.343) | -10.19 (10.836) | -10.49 (12.803)
  Hour 3 | -9.24 (13.445) | -9.90 (11.353) | -9.28 (11.828)
  Hour 4 | -6.86 (13.397) | -8.65 (11.740) | -9.80 (12.802)
  Hour 5 | -5.27 (14.782) | -10.79 (12.123) | -8.54 (15.816)
  Hour 6 | -7.83 (12.628) | -11.47 (13.154) | -5.55 (14.870)
  Hour 7 | -7.15 (13.876) | -9.13 (12.990) | -6.23 (14.911)
  Hour 8 | -8.00 (11.858) | -8.90 (11.220) | -7.44 (13.863)
  Hour 9 | -8.88 (8.732) | -9.56 (12.309) | -6.83 (13.290)
  Hour 10 | -6.89 (10.063) | -8.14 (11.244) | -7.07 (13.808)
  Hour 11 | -5.22 (12.401) | -8.69 (12.989) | -5.41 (12.983)
  Hour 12 | -402 (13.637) | -7.39 (13.722) | -5.64 (12.158)
  Hour 13 | -6.84 (12.616) | -6.33 (10.802) | -6.69 (14.822)
  Hour 14 | -4.34 (12.057) | -6.73 (11.751) | -3.97 (14.844)
  Hour 15 | -4.53 (13.244) | -5.51 (10.473) | -3.85 (11.421)
  Hour 16 | -3.91 (11.469) | -7.20 (10.179) | -2.60 (11.997)
  Hour 17 | -6.68 (11.774) | -7.21 (10.460) | -4.43 (11.789)
  Hour 18 | -5.87 (12.152) | -6.94 (10.904) | -6.36 (11.225)
  Hour 19 | -5.32 (9.200) | -7.61 (11.841) | -3.94 (11.700)
  Hour 20 | -5.17 (16.028) | -10.45 (10.969) | -3.06 (10.965)
  Hour 21 | -6.97 (12.581) | -9.44 (9.303) | -6.33 (12.257)
  Hour 22 | -7.57 (11.891) | -11.37 (10.507) | -6.61 (12.324)
  Hour 23 | -6.12 (13.266) | -9.95 (10.374) | -9.89 (15.553)
  Hour 24 | -5.23 (10.793) | -8.62 (10.066) | -7.19 (10.504)

8. Secondary Outcome: Sub-group Analysis for Change From Baseline in Mean Ambulatory Systolic Blood Pressure in Non-dippers.
Description: as for outcome 6
Time Frame: baseline, 8 weeks
Population: A subset of participants, who participated in ambulatory blood pressure monitoring, was analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 165 | 156 | 148
mmHg
  Hour 1 | -11.29 (15.196) | -10.38 (15.257) | -9.37 (16.751)
  Hour 2 | -10.51 (16.652) | -11.07 (17.183) | -10.26 (16.202)
  Hour 3 | -10.03 (15.654) | -9.82 (18.755) | -9.10 (17.448)
  Hour 4 | -8.79 (17.070) | -5.77 (17.588) | -7.55 (19.225)
  Hour 5 | -7.84 (17.290) | -8.15 (16.984) | -6.40 (19.817)
  Hour 6 | -8.71 (16.700) | -7.77 (17.722) | -6.51 (19.439)
  Hour 7 | -9.07 (17.599) | -8.27 (19.157) | -6.93 (17.751)
  Hour 8 | -11.07 (16.115) | -8.30 (16.824) | -6.36 (18.156)
  Hour 9 | -10.31 (16.749) | -10.65 (15.636) | -8.70 (18.304)
  Hour 10 | -11.48 (16.782) | -10.68 (17.256) | -7.55 (18.870)
  Hour 11 | -10.01 (15.182) | -8.96 (19.195) | -9.49 (17.537)
  Hour 12 | -12.37 (15.745) | -11.55 (18.456) | -8.25 (17.806)
  Hour 13 | -13.49 (17.706) | 10.64 (19.736) | -9.82 (18.908)
  Hour 14 | -13.20 (16.747) | -13.34 (18.467) | -10.24 (17.972)
  Hour 15 | -14.01 (17.729) | -11.95 (16.789) | -12.62 (16.855)
  Hour 16 | -15.15 (15.683) | -14.04 (15.090) | -12.52 (15.137)
  Hour 17 | -14.00 (16.145) | -14.71 (16.069) | -11.71 (17.849)
  Hour 18 | -15.93 (16.180) | -15.37 (14.999) | -9.97 (17.116)
  Hour 19 | -16.45 (16.800) | -16.04 (15.968) | -10.37 (15.684)
  Hour 20 | -15.29 (16.220) | -14.20 (16.727) | -10.90 (15.129)
  Hour 21 | -14.10 (15.413) | -15.26 (17.307) | -10.52 (16.818)
  Hour 22 | -13.97 (15.504) | -12.79 (14.252) | -10.67 (17.877)
  Hour 23 | -11.91 (15.622) | -9.55 (17.616) | -10.77 (15.363)
  Hour 24 | -13.07 (15.572) | -11.81 (16.006) | -7.57 (15.992)

9. Secondary Outcome: Sub-group Analysis for Change From Baseline in Mean Ambulatory Diastolic Blood Pressure in Non-dippers.
Description: as for outcome 6
Time Frame: baseline, 8 weeks
Population: A subset of participants, who participated in ambulatory blood pressure monitoring, was analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 165 | 156 | 148
mmHg
  Hour 1 | -5.93 (9.153) | -6.57 (10.350) | -4.57 (10.648)
  Hour 2 | -5.41 (10.593) | -551 (11.655) | -5.49 (11.892)
  Hour 3 | -3.95 (11.359) | -4.20 (12.472) | -4.44 (12.069)
  Hour 4 | -3.68 (13.107) | -3.53 (11.966) | -4.70 (12.290)
  Hour 5 | -3.53 (13.159) | -3.14 (12.208) | -3.81 (13.309)
  Hour 6 | -4.10 (12.180) | -3.55 (10.888) | -2.94 (13.162)
  Hour 7 | -4.85 (12.321) | -3.31 (12.281) | -2.71 (13.000)
  Hour 8 | -6.07 (11.764) | -2.22 (11.449) | -3.44 (12.022)
  Hour 9 | -4.34 (11.489) | -4.78 (10.645) | -4.54 (12.454)
  Hour 10 | -5.53 (10.639) | -4.48 (10.549) | -3.57 (12.906)
  Hour 11 | -4.53 (10.520) | -4.10 (11.889) | -5.51 (13.254)
  Hour 12 | -5.43 (10.795) | -4.42 (11.973) | -4.50 (11.743)
  Hour 13 | -5.57 (12.269) | -5.01 (13.670) | -6.04 (12.832)
  Hour 14 | -6.18 (12.291) | -5.91 (12.409) | -5.26 (12.249)
  Hour 15 | -7.29 (12.351) | -5.95 (11.443) | -7.52 (12.395)
  Hour 16 | -7.68 (12.231) | -7.26 (10.726) | -6.96 (11.524)
  Hour 17 | -7.28 (12.097) | -7.84 (11.479) | -6.14 (12.302)
  Hour 18 | -8.38 (11.421) | -8.81 (10.385) | -5.28 (12.401)
  Hour 19 | -9.02 (11.661) | -8.77 (10.560) | -5.20 (11.211)
  Hour 20 | -8.92 (11.687) | -7.12 (10.020) | -5.80 (11.234)
  Hour 21 | -8.05 (10.480) | -7.24 (12.056) | -6.49 (12.078)
  Hour 22 | -7.16 (10.060) | -6.55 (8.317) | -5.65 (11.711)
  Hour 23 | -6.34 (10.752) | -5.19 (11.593) | -6.26 (9.552)
  Hour 24 | -5.86 (9.930) | -6.05 (9.926) | -4.96 (9.716)

10. Secondary Outcome: Number of Patients Achieving Successful Blood Pressure Control
Description: Successful blood pressure control is defined as msSBP <140 mmHg and msDBP <90 mmHg.
Time Frame: 8 weeks
Population: Participants from the full analysis set (FAS), who had both baseline and endpoint, were included in the analysis. The FAS included all participants who received study medication and had post baseline BP assessments.
Measure: Number; unit: Number of participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 477 | 469 | 481
Number of participants | 256 | 270 | 235

11. Secondary Outcome: Change From Baseline in Ambulatory Pulse Pressure
Description: Ambulatory pulse pressure (PP) is calculated by hourly ambulatory SBP and hourly ambulatory DBP over a 24-hour period.
Time Frame: baseline, 8 weeks
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 184 | 182
mmHg | -5.78 (0.23) | -5.98 (0.23) | -4.58 (0.23)

12. Secondary Outcome: Number of Responders
Description: Responders are patients with msSBP response (<140 mmHg or ≥20 mmHg reduction from baseline) and msDBP response (<90 mmHg or ≥10 mmHg reduction from baseline)
Time Frame: baseline, 8 weeks
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 477 | 469 | 481
Participants | 312 | 314 | 290

13. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events, and Death as Assessment of Safety and Tolerability
Description: Participants were monitored for adverse events, serious adverse events and deaths throughout the study.
Time Frame: baseline, 8 weeks
Population: Safety Set (SAF): All patients who received at least one dose of double-blind trial medication. Patients were analyzed according to the treatment they received.
Measure: Number; unit: Participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 478 | 472 | 484
Participants
  Adverse events (non-serious and serious | 143 | 132 | 134
  Serious adverse events | 5 | 3 | 6
  Deaths | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Serious Adverse Events (participants affected / at risk) | 5/478 | 3/472 | 6/484
Other Adverse Events (participants affected / at risk) | 66/478 | 63/472 | 66/484
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 200 mg (N=478) | LCZ696 400 mg (N=472) | Olmesartan 20 mg (N=484)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1
BILE DUCT STONE (Hepatobiliary disorders) | 1 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0
DENGUE FEVER (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 200 mg (N=478) | LCZ696 400 mg (N=472) | Olmesartan 20 mg (N=484)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 15 | 5 | 8
BLOOD GLUCOSE INCREASED (Investigations) | 5 | 10 | 13
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 16 | 22 | 21
HYPERURICAEMIA (Metabolism and nutrition disorders) | 14 | 13 | 16
DIZZINESS (Nervous system disorders) | 8 | 11 | 3
HEADACHE (Nervous system disorders) | 6 | 4 | 10
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.